CLINICAL TRIAL: NCT00003783
Title: ALinC 17: Continuous Intensification for Very High Risk Acute Lymphocytic Leukemia (A.L.L.): A Pediatric Oncology Group Pilot Study
Brief Title: Combination Chemotherapy in Treating Children With Very High Risk Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9806; POG-9806 (Other: Pediatric Oncology Group); CDR0000066915 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; Etoposide; Idarubicin; Leucovorin; Mercaptopurine; Methotrexate; Prednisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complete Response and no CNS 3 (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: etoposide; Drug: idarubicin; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy
- Complete Response and CNS 3 (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: etoposide; Drug: idarubicin; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: G-CSF
Drug: asparaginase
  Other Names: E. coli; Elspar; NSC #109229
Drug: cyclophosphamide
  Other Names: CTX; Cytoxan; NSC #026271
Drug: cytarabine
  Other Names: cytosine arabinoside; Ara-C; Cytosar; NSC #063878
Drug: daunorubicin hydrochloride
  Other Names: daunomycin; DNR; Cerubidine; NSC #82151
Drug: dexamethasone
  Other Names: Decadron; NSC #034521
Drug: etoposide
  Other Names: VP-16; VePesid; NSC #141540
Drug: idarubicin
  Other Names: 4-demethoxydaunorubicin; Idamycin; NSC #256439
Drug: leucovorin calcium
  Other Names: LCV; Wellcovorin; citrovorum factor; folinic acid; NSC #003590
Drug: mercaptopurine
  Other Names: 6-MP; Purinethol; NSC #000755
Drug: methotrexate
  Other Names: MTX; amethopterin; NSC #000740; IND #4291
Drug: prednisone
  Other Names: Deltasone; Meticorten; Liquid Pred; NSC #010023
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC #067574
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug and combining drugs in different ways may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy in treating children who have very high risk acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of administering a new combination of agents during postinduction consolidation therapy in children with very high risk acute lymphocytic leukemia (VHR-ALL). II. Assess the tolerance of patients in remission of VHR-ALL for postconsolidation therapy with continuous intensification.

OUTLINE: Patients receive induction therapy on weeks 1-4. This consists of oral prednisone three times a day on days 1-28; vincristine IV on days 1, 8, 15, and 22; daunorubicin IV on days 8, 15, and 22; and asparaginase IM on days 2, 5, 8, 12, 15, and 19. Patients also receive methotrexate intrathecally (IT) on days 1 and 8. Patients with CNS 2 and 3 disease also receive methotrexate IT on days 15 and 22. Patients who achieve M2 bone marrow on day 29 receive oral prednisone three times a day on days 29-42; vincristine IV and daunorubicin IV over 15 minutes on days 29 and 36; and asparaginase IM on days 29, 32, 36, and 39. If bone marrow is M3 on day 29 or M2 or M3 on day 43, then patient is off study. Patients proceed to consolidation therapy on weeks 5-25. This consists of high dose methotrexate IV over 24 hours on weeks 6, 8, 16, and 18, followed by leucovorin calcium IV or orally every 6 hours for 5 doses; oral mercaptopurine on weeks 6-9 and 16-19; cytarabine IV over 6 hours followed by idarubicin IV over 15 minutes for 4 days; and filgrastim (G-CSF) subcutaneously (SQ) beginning on day 5 and continuing for about 10-14 days on weeks 10 and 20. Patients receive etoposide IV over 1 hour followed by cyclophosphamide IV over 10 minutes for 5 days and G-CSF SQ beginning on day 6 for 10-14 days on weeks 13 and 23. Methotrexate IT is administered on weeks 6, 8, 13, 16, 18, and 23. Patients then proceed to continuous intensification therapy during weeks 26-61. Patients receive vincristine IV, daunorubicin IV, and methotrexate IT on day 1, and oral dexamethasone twice a day on days 1-7 on weeks 26, 32, 38, 44, 50, and 56. Patients also receive high dose cytarabine IV over 1 hour, every 12 hours, for 4 doses, followed by asparaginase IM 3 hours after the last dose of cytarabine, on weeks 27, 33, 39, 45, 51, and 57. Oral mercaptopurine and methotrexate IM are administered on day 1 during weeks 29, 31, 35, 37, 41, 43, 47, 49, 53, 55, 59, and 61. Patients receive etoposide IV over 1-2 hours followed by cyclophosphamide IV during weeks 30, 36, 42, 48, 54, and 60. Patients then proceed to continuation therapy during weeks 62-126. Vincristine IV and cyclophosphamide IV are administered on weeks 62-65, 70-73, 78-81, 86-89, 94-97, 102-105, 110-113, and 118-121. Patients also receive oral dexamethasone twice a day for 7 days on weeks 62, 70, 78, 86, 94, 102, 110, and 118, and cytarabine IV on weeks 63, 65, 71, 73, 79, 81, 87, 89, 95, 97, 103, 105, 111, 113, 119, and 121. Oral mercaptopurine is administered daily during weeks 66-69, 74-77, 82-85, 90-93, 98-101, 106-109, 114-117, and 122-125 and methotrexate IM on weeks 66-69, 74-77, 82-85, 90-93, 98-101, 106-109, 114-117, and 122-125. Methotrexate IT is administered during weeks 62, 70, 78, 86, 94, 102, 110, and 118. Patients who are CNS 3 at diagnosis receive whole brain irradiation beginning at week 62 along with the first course of continuation therapy. These patients do not receive any methotrexate IT after week 62. Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, every 6 months for 1 year, then annually thereafter.

PROJECTED ACCRUAL: A total of 38 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed B-cell precursor acute lymphocytic leukemia No L3 morphology Very poor prognosis CNS 3 (blasts and WBC greater than 5 microliters) OR Must meet all of the following criteria: No simultaneous trisomy 4 and 10 DNA index no greater than 1.16 (if FISH 4 and 10 unsatisfactory) No TEL-AML1 [t(12;21)] Meets at least 1 of the following: Has MLL (11q23) and/or BCR-ABL [t(9;22)] WBC greater than 100,000/mm3 Age over 12 (boys) or 16 (girls) OR Boys Girls WBC 8 12 greater than 80,000/mm3 9 13 greater than 60,000/mm3 10 14 greater than 40,000/mm3 11 15 greater than 20,000/mm3 Concurrent registration on stratum 6 of POG-9400 before 11/15/1999 OR Concurrent registration on stratum 4 of POG-9900 after 11/15/1999 Concurrent registration on POG-9201, POG-9705, or POG-9806 unless ineligible

PATIENT CHARACTERISTICS: Age: Children Performance status: Not specified Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 1999-03; Primary Completion 2002-11 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility of delivering a new combination of agents during a 20 week post-induction consolidation phase | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William P. Bowman, MD, Study Chair — Cook Children's Medical Center - Fort Worth
Locations (58):
- United States (51):
  - Arizona Cancer Center, Tucson, Arizona
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Portland, Maine
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Roanoke Community Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Medical School, Charleston Division, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland